CLINICAL TRIAL: NCT01548833
Title: Randomized Cross-Over Evaluation of Silicone Hydrogel Daily Disposable Soft Contact Lenses
Brief Title: Pre-Lens Tear Film Performance of Silicone Hydrogel Daily Disposable Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Collaborators: Aston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: A00924
Record Dates: First submitted 2012-03-06; First posted 2012-03-08 (Estimated); Results first posted 2013-06-24 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Myopia
Keywords: Myopia; Contact Lenses
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dailies Total 1 (Experimental): Delefilcon A, followed by narafilcon A and filcon II 3 in randomized order. Each product worn for 1 week in a daily wear, daily disposable manner.
  Interventions: Device: Delefilcon A contact lens; Device: Narafilcon A contact lens; Device: Filcon II 3 contact lens
- TruEye (Active Comparator): Narafilcon A, followed by delefilcon A and filcon II 3 in randomized order. Each product worn for 1 week in a daily wear, daily disposable manner.
  Interventions: Device: Delefilcon A contact lens; Device: Narafilcon A contact lens; Device: Filcon II 3 contact lens
- Clariti (Active Comparator): Filcon II 3, followed by narafilcon A and delefilcon A in randomized order. Each product worn for 1 week in a daily wear, daily disposable manner.
  Interventions: Device: Delefilcon A contact lens; Device: Narafilcon A contact lens; Device: Filcon II 3 contact lens

INTERVENTIONS:
Device: Delefilcon A contact lens — Silicone hydrogel contact lens for single use, daily disposable wear.
  Other Names: DAILIES® TOTAL1™
Device: Narafilcon A contact lens — Silicone hydrogel contact lens for single use, daily disposable wear.
  Other Names: 1-DAY ACUVUE® TRUEYE™
Device: Filcon II 3 contact lens — Silicone hydrogel contact lens for single use, daily disposable wear
  Other Names: Clariti™ 1-day

SUMMARY:
The purpose of this study was to compare the pre-lens tear film stability of DAILIES TOTAL1® silicone hydrogel daily disposable contact lenses with that of two other silicone hydrogel daily disposable contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Be of legal age of consent and sign written Informed Consent document, or if under legal age, have written consent of parent or guardian to participate.
* Require vision correction in both eyes.
* Wear either daily disposable contact lenses or weekly/monthly replacement contact lenses in powers between -0.50 and -10.00 diopters, cylinder ≤0.75 diopter, no ADD correction.
* Wear habitual contact lenses an average of 12-14 hours per day, at least 5 days per week.
* Willing and able to wear study contact lenses 16 hours per day.
* Able to achieve visual acuity of at least 6/7.5 in each eye with study lenses.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Currently wearing DAILIES TOTAL1®, 1-DAY ACUVUE® TRUEYE™, or Clariti™ 1day contact lenses.
* Require monovision correction.
* Any systemic or ocular disease or disorder (refractive disorder allowed and dry eye permitted), complicating factors, or structural abnormality that would negatively affect the conduct or outcome of the study.
* Ocular surgery/trauma within the last 6 months.
* Topical or systemic antibiotic use within 7 days of enrollment.
* Topical ocular or systemic corticosteroid use within 14 days of enrollment.
* Pregnant and nursing women.
* Participation in any other ophthalmic drug or device clinical trial within 30 days of enrollment.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jami Kern, PhD, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one study center in the United Kingdom.
Pre-assignment Details: This reporting group includes all enrolled participants.
Groups:
- Overall: All enrolled participants
Period: Overall Study
Arm/Group | Overall
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Overall: DT1, TruEye, and Clariti contact lenses worn in randomized, cross-over fashion for one week each
Arm/Group | Overall
Number analyzed (Participants) | 39
Age Continuous [Mean (Standard Deviation); unit: years] | 22.1 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 18
Region of Enrollment [Number; unit: participants]
  United Kingdom | 39

OUTCOME MEASURES:

1. Primary Outcome: Pre-Lens Non-Invasive Tear Break-Up Time (PL-NITBUT)
Description: The pre-lens tear film is the layer of tears located on top of the contact lens (i.e., between the eye lid and the contact lens). The time required for a dry spot to appear on the corneal surface after blinking is referred to as the tear film break-up time. Circular images were projected onto the corneal surface using a CA-1000 topographer, and the tear film reflection was observed on a 30-inch flat panel monitor. PL-NITBUT was recorded at the first sign of image distortion. Three measurements were taken and averaged together. A higher number represents a longer tear film break up time.
Time Frame: Day 7, 16 hours after lens insertion
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Dailies Total 1: Delefilcon A contact lenses worn for one week in a daily wear, daily disposable manner.
- TruEye: Narafilcon A contact lenses worn for one week in a daily wear, daily disposable manner.
- Clariti: Filcon II 3 contact lenses worn for one week in a daily wear, daily disposable manner.
Arm/Group | Dailies Total 1 | TruEye | Clariti
Number analyzed (Participants) | 39 | 39 | 39
seconds | 13.56 (3.7759121) | 12.0 (2.9676727) | 11.86 (3.5982819)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the trial.
Arm/Group | Dailies Total 1 | TruEye | Clariti
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 0/39 | 0/39 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.